CLINICAL TRIAL: NCT01584713
Title: A Phase II Clinical Trial to Study the Feasibility and Safety of Stromal Vascular Derived From Adipose Tissue for the Treatment of Enterocutaneous Fistula
Brief Title: Stromal Vascular Fraction (SVF) for Treatment of Enterocutaneous Fistula (HULPUTC)
Acronym: HULPUTC
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto de Investigación Hospital Universitario La Paz (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EC10-345; 2010-024308-82 (EudraCT Number)
Record Dates: First submitted 2012-02-26; First posted 2012-04-25 (Estimated); Last update posted 2012-04-25 (Estimated); Status verified 2012-04

CONDITIONS: Enterocutaneous Fistula
Keywords: Enterocutaneous fistula; Adipose Derived Stem Cells
MeSH Terms: conditions — Intestinal Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Adipose derived Stem Cells (Experimental)
  Interventions: Drug: Adipose-derived stem cells without expanded

INTERVENTIONS:
Drug: Adipose-derived stem cells without expanded — Administration will be intralesional injection of cells suspension. They will be placed into fistula walls
  Other Names: Non applicable

SUMMARY:
The purpose of this study is to determine safety of Stromal Vascular Fraction (SVF) for the treatment of enterocutaneous fistula.

DETAILED DESCRIPTION:
SF-12 Test

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Enterocutaneous fistula
* Men and women over 18 years old. Good general state of health according to the findings of the clinical history and the physical examination

Exclusion Criteria:

* Presence of severe proctitis or dominant active luminal disease requiring immediately therapy
* Patients with an abscess unless a complete toilet of the area with drainage of the collections and the absence of abscess and other collections is confirmed prior to treatment start
* Patients with a history of abuse of alcohol or other addictive substances in the 6 months prior to inclusion
* Patients with malignant tumor, except for basal cell or cutaneous squamous cell carcinoma, or patients with a prior history of malignant tumors, unless the neoplastic disease has been in remission for the previous 5 years
* Patients with cardiopulmonary disease which, in opinion of the investigator, in unstable or sufficiently serious to exclude the patient from the study.
* Patients with any type of medical or psychiatric disease which, in the opinion of the investigator, could be grounds for exclusion from study
* Patients with congenital or acquired immunodeficiencies. HIV, HBV, HCV or treponema infection, whether active or latent
* Patients who have suffering major surgery or severe trauma in the prior 6 months
* Pregnant or breastfeeding women
* Patients currently receiving, or having received within 1 month prior to enrollment into this clinical trial, any investigational drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2011-12; Primary Completion 2012-07 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Safety of treatment of treated enterocutaneous fistulae. Percentage of treated subjects with closed fistulae | 16 weeks
  Safety by analyzing the number of adverse effects associated with experimental treatment.

SECONDARY OUTCOMES:
quality of life test | 16 week
  Test SF 12 of quality of life
First efficacy data | 16 weeks
  Fistula closure by radiology

CONTACTS AND LOCATIONS:
Overall Officials: Mariano Garcia-Arranz, Doctor, Principal Investigator — Fundacion para la Investigacion Biomedica del Hospital Universitario la Paz
Locations (1):
- Hospital Universitario La Paz, Madrid, Madrid, Spain

REFERENCES:
- [Background] Garcia-Olmo D, Garcia-Arranz M, Herreros D, Pascual I, Peiro C, Rodriguez-Montes JA. A phase I clinical trial of the treatment of Crohn's fistula by adipose mesenchymal stem cell transplantation. Dis Colon Rectum. 2005 Jul;48(7):1416-23. doi: 10.1007/s10350-005-0052-6. PMID 15933795
- [Background] Garcia-Olmo D, Garcia-Arranz M, Herreros Marcos D, Pascual Miguelañez I. Fibrina y terapia celular en el tratamiento de la patología fistulosa en la enfermedad de Crohn. Protocolo y resultados de un ensayo clínico en fase I. Rev Esp Enferm Dig 2005. 97(Supl. II):51-54.)
- [Background] Herreros Marcos D, Garcia-Arranz M, Pascual Miguelañez I, Garcia-Olmo D. THE ROLE OF STEM CELLS IN SUPPURATIVE ENVIROMENTS. Experimental Dermatology 2006, 15 (6): 482.
- [Background] García Olmo D, Trébol J, Herreros D, Garcia-Arranz M, Gonzalez M. TREATMENT OF FISTULAS USING ADIPOSE-DERIVED STEM CELLS. En: García Olmo D, García-Verdugo JM, Alemany J, Gonzalez M, Gutierrez-Fuentes JA. CELL THERAPHY .2008 Ed. Mac Graw Hill. Madrid 2007
- [Background] Alvarez PD, Garcia-Arranz M, Georgiev-Hristov T, Garcia-Olmo D. A new bronchoscopic treatment of tracheomediastinal fistula using autologous adipose-derived stem cells. Thorax. 2008 Apr;63(4):374-6. doi: 10.1136/thx.2007.083857. PMID 18364447
- [Background] Garcia-Olmo D, Garcia-Arranz M, Herreros D. Expanded adipose-derived stem cells for the treatment of complex perianal fistula including Crohn's disease. Expert Opin Biol Ther. 2008 Sep;8(9):1417-23. doi: 10.1517/14712598.8.9.1417. PMID 18694359
- [Background] Pascual I, de Miguel GF, Gomez-Pinedo UA, de Miguel F, Arranz MG, Garcia-Olmo D. Adipose-derived mesenchymal stem cells in biosutures do not improve healing of experimental colonic anastomoses. Br J Surg. 2008 Sep;95(9):1180-4. doi: 10.1002/bjs.6242. PMID 18690635
- [Background] Vilalta M, Degano IR, Bago J, Gould D, Santos M, Garcia-Arranz M, Ayats R, Fuster C, Chernajovsky Y, Garcia-Olmo D, Rubio N, Blanco J. Biodistribution, long-term survival, and safety of human adipose tissue-derived mesenchymal stem cells transplanted in nude mice by high sensitivity non-invasive bioluminescence imaging. Stem Cells Dev. 2008 Oct;17(5):993-1003. doi: 10.1089/scd.2007.0201. PMID 18537463
- [Background] Garcia-Olmo D, Herreros D, Pascual I, Pascual JA, Del-Valle E, Zorrilla J, De-La-Quintana P, Garcia-Arranz M, Pascual M. Expanded adipose-derived stem cells for the treatment of complex perianal fistula: a phase II clinical trial. Dis Colon Rectum. 2009 Jan;52(1):79-86. doi: 10.1007/DCR.0b013e3181973487. PMID 19273960
- [Background] Garcia-Olmo, D; Guadalajara, H; Trebol, J, García-Arranz M. Expanded Adipose-Derived Stem Cells for the Treatment of Complex Perianal Fistula. HUMAN GENE THERAPY 2009. 20 (9):1028-1028
- [Background] Trebol, J; Garcia-Arranz, M; Georgiev-Hristov, T, et al. Cell Therapy for Enterocutaneous Fistula Associated with Crohn's Disease: A Clinical and Biological Comparison of Protocols With and Without Cell Expansion. HUMAN GENE THERAPY 2009. 20 (9): 1045-1045
- [Background] Garcia-Gomez, I; Olmedillas, S; Garcia-Arranz, M, et al. Adipose-Derived Stem Cells Reduce Abdominal Adhesion Formation in a Rat Experimental Model. HUMAN GENE THERAPY 2009. 20 (9): 1047-1047
- [Background] Georgiev-Hristov, T; Garcia-Olmo, D; Alvarez, PDA, et al. Use of Surgical Sutures Enriched with Adipose-Derived Stem Cells for Tracheal Anastomosis in Rats. HUMAN GENE THERAPY 2009. 20 (9): 1074-1075
- [Background] Vicente, A; Vazquez, MN; Entrena, A, Gqarcía-Arranz M,et al. BMP-4 Regulates the Expansion and Survival of Human Adipose Mesenchymal Cells. HUMAN GENE THERAPY .2009. 20 (9):1080-1081
- [Background] Garcia-Olmo D, Herreros D, Pascual M, Pascual I, De-La-Quintana P, Trebol J, Garcia-Arranz M. Treatment of enterocutaneous fistula in Crohn's Disease with adipose-derived stem cells: a comparison of protocols with and without cell expansion. Int J Colorectal Dis. 2009 Jan;24(1):27-30. doi: 10.1007/s00384-008-0559-0. Epub 2008 Aug 12. PMID 18696086
- [Background] Garcia-Olmo D, Herreros D, De-La-Quintana P, Guadalajara H, Trebol J, Georgiev-Hristov T, Garcia-Arranz M. Adipose-derived stem cells in Crohn's rectovaginal fistula. Case Rep Med. 2010;2010:961758. doi: 10.1155/2010/961758. Epub 2010 Mar 7. PMID 20224798
- [Background] Pascual I, Fernandez de Miguel G, Garcia Arranz M, Garcia-Olmo D. Biosutures improve healing of experimental weak colonic anastomoses. Int J Colorectal Dis. 2010 Dec;25(12):1447-51. doi: 10.1007/s00384-010-0952-3. Epub 2010 Jun 11. PMID 20544210
- [Background] Garcia-Arranz M, Gomez-Pinedo U, Hardisson D, Herreros D, Guadalajara H, Garcia-Gomez I, Garcia-Verdugo JM, Garcia-Olmo D. Histopathological analysis of human specimens removed from the injection area of expanded adipose-derived stem cells. Histopathology. 2010 Jun;56(7):979-82. doi: 10.1111/j.1365-2559.2010.03573.x. No abstract available. PMID 20636801
- [Background] Garcia-Gomez I, Elvira G, Zapata AG, Lamana ML, Ramirez M, Castro JG, Arranz MG, Vicente A, Bueren J, Garcia-Olmo D. Mesenchymal stem cells: biological properties and clinical applications. Expert Opin Biol Ther. 2010 Oct;10(10):1453-68. doi: 10.1517/14712598.2010.519333. PMID 20831449
- [Background] Vicente Lopez MA, Vazquez Garcia MN, Entrena A, Olmedillas Lopez S, Garcia-Arranz M, Garcia-Olmo D, Zapata A. Low doses of bone morphogenetic protein 4 increase the survival of human adipose-derived stem cells maintaining their stemness and multipotency. Stem Cells Dev. 2011 Jun;20(6):1011-9. doi: 10.1089/scd.2010.0355. Epub 2010 Nov 4. PMID 20846028
- [Background] Trebol Lopez J, Georgiev Hristov T, Garcia-Arranz M, Garcia-Olmo D. Stem cell therapy for digestive tract diseases: current state and future perspectives. Stem Cells Dev. 2011 Jul;20(7):1113-29. doi: 10.1089/scd.2010.0277. Epub 2011 Feb 17. PMID 21187000
- [Background] Garcia-Olmo D, Garcia-Arranz M. [Cells for curing. From the heart to everything]. An Pediatr (Barc). 2011 Apr;74(4):215-7. doi: 10.1016/j.anpedi.2011.02.021. No abstract available. Spanish. PMID 21459345
- [Background] Garcia-Olmo D, Herreros D, Guadalajara H, Trebol J, Georgiev T, García-Arranz M.Adipose Derived Stem Cell for Treatment of Crohn´s fistula. Histology and Histopathology. 2011; 26(ss1):356